CLINICAL TRIAL: NCT00662532
Title: Multi-Center Phase 3 Trial of Minocycline HCl 1mg Microspheres for the Use in Subjects With Peri-Implantitis
Brief Title: Antibiotic Study for Dental Implants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OraPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP-P-5265-1
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Periodontitis
Keywords: Peri-implantitis; antibiotic
MeSH Terms: conditions — Periodontitis; Peri-Implantitis | interventions — Minocycline; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline HCl (Experimental): 1 mg microspheres of minocycline hydrochloride
  Interventions: Drug: Minocycline HCl
- No Intervention (No Intervention): Control group receiving no drug intervention

INTERVENTIONS:
Drug: Minocycline HCl — 1mg microspheres for professional subgingival administration into periodontal pockets two times throughout the duration of the trial
  Other Names: antibiotic
  Arms: Minocycline HCl

SUMMARY:
This study is for people at least 21 years old who have signs of problems, like swollen gums and shrinking bones, by dental implants.

DETAILED DESCRIPTION:
At Visit 1, the dentist will:

* do an oral exam
* ask some questions
* decide if the person qualifies for being in the study
* make an appointment for Visit 2 if they qualify

At Visit 2 (Baseline), the dentist will:

* do a special cleaning of the implants
* examine the whole mouth
* collect some fluid
* take x-rays
* put the people into one of two groups (taking into account whether or not they smoke)

  1. one group will have the study antibiotic put on all the areas in their mouth with gum problems
  2. the other group will not receive the antibiotic At Visit 3 (about a month later), only fluid samples will be collected.

At Visit 4 (about 3 months later), the dentist will:

* collect fluid samples
* examine the whole mouth
* apply the antibiotic again for people in that group

At Visit 5 (about 6 months later), the dentist will:

* collect fluid samples
* examine the whole mouth
* take x-rays

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and good general health
* appropriately documented Informed Consent
* willing to adhere to the study schedule, prohibitions and restrictions specified in the protocol
* female subjects must meet the pregnancy and contraceptive requirements
* must have oral health appropriate for study inclusion

Exclusion Criteria:

* oral health inappropriate for study inclusion
* females self-reporting pregnancy or lactation, or having a positive urine pregnancy result
* reporting any of the following conditions:
* allergy to a tetracycline-class drug
* systemic medical conditions requiring antibiotic prophylaxis prior to invasive dental procedures
* active systemic infectious disease such as hepatitis, human immunodeficiency virus (HIV) or tuberculosis
* diagnosed with clinically significant or unstable organic disease, or compromised healing potential, heart murmurs, histories of rheumatic fever, valvular disease or prosthetic joint replacement
* participation in a dental clinical trial or use of an investigational drug within 30 days of enrollment
* employees of the Investigator or study center, with direct involvement in the proposed study or other studies, as well as family members of the employees or the Investigator
* anyone who the investigator determines should not be included in the study for any reason that could compromise safety or the analysis of study results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — OraPharma
Locations (4):
- United States (4):
  - JJCPPW Investigational Site, Aurora, Colorado
  - JJCPPW Investigational Site, Ann Arbor, Michigan
  - JJCPPW Investigational Site, Hazlet, New Jersey
  - JJCPPW Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline HCl | No Intervention
Started | 22 | 22
Completed | 22 | 20
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline HCl | No Intervention | Total
Number analyzed (Participants) | 22 | 22 | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 67.59 (12.37) | 66.05 (10.97) | 66.82 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall PD Reduction
Description: Mean reduction of probing depth (PD) of qualified implant sites is derived by calculating the change of PD per qualified implant site (PD at baseline minus PD at post-baseline), and then averaging the site-specific PD changes per subject
Time Frame: Baseline to Day 180
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Minocycline HCl | No Intervention
Number analyzed (Participants) | 22 | 22
mm | 1.25 (0.63) | 0.66 (0.63)

2. Secondary Outcome: Initial PD Reduction
Description: as for outcome 1
Time Frame: Baseline to Day 90
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Minocycline HCl | No Intervention
Number analyzed (Participants) | 22 | 22
mm | 1.02 (0.63) | 0.49 (0.58)

3. Secondary Outcome: BOP Percent Reduction From Baseline
Description: Bleeding on Probing (BOP) percentage is calculated as the number of implant sites with bleeding divided by the number of implant sites per subject times 100% at each visit; reduction of BOP percentage is the BOP percentage at baseline minus the BOP percentage post-baseline
Time Frame: at Day 90 and Day 180
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Minocycline HCl | No Intervention
Number analyzed (Participants) | 22 | 22
Percentage of Participants
  Day 90 | 42.17 (38.27) | 22.53 (31.36)
  Day 180 | 60.75 (32.19) | 32.86 (41.35)

ADVERSE EVENTS:
Time Frame: 180 Days
Description: Adverse Events were a primary outcome measure, so we have used a 1% reporting threshold, rather than the standard 5%
Arm/Group | Minocycline HCl | No Intervention
Serious Adverse Events (participants affected / at risk) | 1/22 | 3/22
Other Adverse Events (participants affected / at risk) | 6/22 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline HCl (N=22) | No Intervention (N=22)
Volvulus (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline HCl (N=22) | No Intervention (N=22)
Tooth Abscess (Infections and infestations) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Bite (Injury, poisoning and procedural complications) | 1 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1
Endodontic Procedure (Surgical and medical procedures) | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 1
Nodule (General disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No